CLINICAL TRIAL: NCT02742948
Title: The Optimal Time for Intravenous Antibiotic Prophylaxis in Elective Cesarean Section: Randomized Comparative Study
Brief Title: The Optimal Time for Intravenous Antibiotic Prophylaxis in Elective Cesarean Section
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, lecturer of obs& gyn, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 821978
Record Dates: First submitted 2016-03-30; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Endometritis
Keywords: elective caesarean section; antibiotics; endometritis
MeSH Terms: conditions — Endometritis | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- preoperative antibiotic group (Active Comparator): 200 women will receive IV ceftriaxone (2g) 60 minutes before skin incision
  Interventions: Drug: ceftriaxone
- early intraoperative antibiotic group (Active Comparator): 200 women will receive IV ceftriaxone (2g) immediately with skin incision
  Interventions: Drug: ceftriaxone
- post cord clamping antibiotic group (Active Comparator): 200 women will receive IV ceftriaxone (2g) immediately after umbilical cord clamping
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone — IV ceftriaxone (2g) will be given to all participants
  Other Names: Rocephin

SUMMARY:
Objective: To determine the optimal time for intravenous antibiotic prophylaxis administration in pregnant women undergoing elective cesarean section to minimize postpartum infectious complication for both the mother & neonate.

Study Design: A randomized comparative study. Setting: The Obstetrics and Gynecology department of Kasr El Aini hospital (Cairo University - Egypt) in the period from April 2016 to September 2016.

Methodology: Six hundred pregnant women aged from 20 to 40 years old with singleton living healthy fetuses undergoing elective lower segment caesarean section (LSCS).They will be randomized into three groups: group A in which 200 women will receive IV ceftriaxone (2g) 60 minutes before skin incision, group B in which 200 women will receive IV ceftriaxone (2g) immediately with skin incision & group C in which 200 women will receive IV ceftriaxone (2g) immediately after umbilical cord clamping. Outcomes include postoperative maternal & fetal infectious morbidity.

DETAILED DESCRIPTION:
Six hundred pregnant women aged from 20 to 40 years old with singleton living healthy fetuses undergoing elective lower segment caesarean section (LSCS); defined as LSCS done before onset of labor pains, will be enrolled in the study. They will be randomized into three groups: group A in which 200 women will receive IV ceftriaxone (2g) 60 minutes before skin incision, group B in which 200 women will receive IV ceftriaxone (2g) immediately with skin incision & group C in which 200 women will receive IV ceftriaxone (2g) immediately after umbilical cord clamping. Randomization will be done using computer generated random numbers.

Another inclusion criterion includes gestational age (GA) more than 37 weeks gestation. Patients on immunosuppressant drugs, received any antibiotic prophylaxis (within 10 days), suffer any chronic illness (e.g. diabetes mellitus or renal disease) or who experienced any obstetric complication in the current pregnancy (e.g. antepartum hemorrhage & rupture of membranes) will be excluded from the study. Additional exclusion criteria include previous history of more than two laparotomies, maternal BMI more than 28 & any maternal febrile illness within 10 days from the procedure. Patients who are known to be allergic to penicillin or cephalosporin will be also excluded (all patients will receive 100 mg of ceftriaxone as a test dose before participation in the current study). The study was approved by the Hospital Ethical Committee. All participants will provide an informed consent after explaining the aim and potential hazards of the study.

For all patients, full history will be taken followed by complete physical examination, obstetric ultrasound & routine preoperative investigations. GA is established by menstrual dates then confirmed by obstetric ultrasound. Spinal anaesthesia will be given for all patients. All cesarean sections will be done by ob/gyn residents under the supervision of senior staff obstetrician using the following technique: Pfannenstiel skin incision, transverse lower uterine segment incision, two-layer closure of the uterine wall, closure of both parietal peritoneum & rectus sheath & skin closure (using prolene 3/0 suture). Primary maternal outcome includes postoperative endometritis (diagnosed if maternal axillary temperature ≥ 38°C for at least 48 hours, uterine tenderness, infected lochia & leukocytosis).Secondary maternal outcomes include wound infection (diagnosed if there is induration, redness, hematoma, seroma or purulent discharge at the incision site) & urinary tract infection (diagnosed if there frequency, dysuria, suprapubic or loin pain & positive urine culture). Prolonged postoperative hospital stay (more than 2 days) will also be recorded. The infectious morbidity evaluation will be done by ob/gyn residents who will be blinded to the study group of the patient. Neonatal outcomes include immediate antibiotic adverse effects (diarrhea & rash), neonatal sepsis (diagnosed by clinical signs, leukocytosis, C-reactive protein& positive blood culture), neonatal intensive care unit (NICU) admission (entailing the length of stay) & neonatal death. All neonates will be examined by an expert neonatologist who will be blinded to study group of the neonate's mother. On discharging all patients, a brief summary about symptoms and signs of the above mentioned infectious & neonatal complications will be given and they will be instructed to contact any of the authors immediately if any happens. Patients will be reexamined after 1 week (skin stitch removal appointment) & 4 weeks (contraception counseling appointment) following the CS.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in singleton living healthy fetuses. gestational age (GA) more than 37 weeks gestation

Exclusion Criteria:

* Patients on immunosuppressant drugs, received any antibiotic prophylaxis (within 10 days), suffer any chronic illness (e.g. diabetes mellitus or renal disease) or who experienced any obstetric complication in the current pregnancy (e.g. antepartum hemorrhage & rupture of membranes). Previous history of more than two laparotomies, maternal BMI more than 28 & any maternal febrile illness within 10 days from the procedure. Patients who are known to be allergic to penicillin or cephalosporin

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
endometritis | up to 4 weeks postoperative
  maternal axillary temperature ≥ 38°C for at least 48 hours, uterine tenderness, infected lochia & leukocytosis.

SECONDARY OUTCOMES:
neonatal immediate side effects | within 24 hours postoperative
  diarrhea & fever
neonatal sepsis | up to 1 week postoperative
  clinical signs, leukocytosis, CRP & positive blood culture
neonatal ICU admission | within 24 hours postoperative
Prolonged hospital stay | 2 days
wound infection | up to 4 weeks postoperative
  induration, redness, hematoma, seroma or purulent discharge at the incision site
urinary tract infection | up to 4 weeks postoperative
  frequency, dysuria, suprapubic or loin pain & positive urine culture.

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz Elsherbini, MD, Principal Investigator — Lecturer of obstetrics & gynaecology - Cairo university